CLINICAL TRIAL: NCT03538548
Title: Predictors of Treatment Outcome in Cognitive-Behavioral Therapy for Cocaine Use
Brief Title: Treatment Outcome in CBT for Cocaine Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard Foltin, Professor of Neurobiology (in Psychiatry) and Research Scientist VII, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7022; 1R01DA035846-01A1 (NIH)
Record Dates: First submitted 2018-04-27; First posted 2018-05-29 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine Abuse; Cocaine Use Disorder; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants receive a standard 12-week course of Cognitive Behavioral Therapy for Relapse Prevention (CBT-RP; Carroll, 1998). The treatment protocol will be implemented over 12 weeks, with two 1-hour sessions per week for the first two weeks and one 1-hour session per week thereafter (i.e., a total of 14 sessions).
  Interventions: Behavioral: CBT-RP

INTERVENTIONS:
Behavioral: CBT-RP — CBT-RP is a time-limited, manual guided intervention that aims to develop behavioral and cognitive skills needed to initiate abstinence and prevent relapse. The treatment will help individuals analyze the decision making process to minimize the influence of more immediate reinforcement, develop cognitive strategies to promote the attainment of longer-term goals, practice behavioral strategies to reduce the influence of socially mediated threats to abstinence, and outline explicit plans for managing situations that threaten their goal of abstinence.

SUMMARY:
Cognitive-behavioral treatments for cocaine abuse could be improved by an increased understanding of factors that predict treatment outcomes. The objective of this protocol is to conduct a study examining the impact of client characteristics on the effects of cognitive-behavioral therapy for cocaine abuse.

DETAILED DESCRIPTION:
Study investigators will recruit treatment-seeking cocaine users (n = 100) from a separate protocol (#6912) who will receive a standard 12-week course of cognitive behavioral therapy for relapse prevention. Using a variety of self-report questionnaires and computer-based tasks, three major domains will be assessed and evaluated as predictors of treatment outcome: (1) impulsivity, (2) motivation to change, and (3) learning style. Measures of these factors will have been obtained in the #6912 protocol. A better understanding of the impact of impulsivity, motivation to change, and learning style on treatment outcome will provide critical information to guide the refinement of CBT for cocaine abuse. For example, the results of this study may help guide the development and introduction of more targeted cognitive remedial strategies or behavioral training components into the framework of evidenced-based practices. These additions may help ameliorate the deleterious effects of specific participant characteristics on the acquisition and implementation of coping skills, which can further improve the efficacy of CBT.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals age 18-60.
2. Currently report using cocaine via the intranasal or smoked route.
3. Be able to give informed consent and comply with study procedures.

Exclusion Criteria:

1. Individuals who meet current (i.e., within the past year) DSM-5 severe Substance Use Disorder (SUD) criteria (defined as the presence of 6 or more symptoms) for drugs other than cocaine, nicotine and caffeine.
2. Individuals who meet current (i.e., within the past year) DSM-5 moderate to severe Major Depressive Disorder criteria (defined as a score of 17 or higher on the Hamilton Depression Rating Scale).
3. Individuals who meet current DSM-5 criteria for any bipolar or psychotic disorder (other than transient psychosis due to drug use), or for all other psychiatric disorders not addressed by other exclusion criteria (e.g., anxiety disorders other than specific phobias, eating disorders, or ADHD) that require medical and/or psychological intervention.
4. Individuals with a neurodevelopmental disorder (e.g., Intellectual Development Disorder, Autism Spectrum Disorder) except ADHD.
5. Individuals with uncorrected visual or auditory deficits, or who cannot adequately read or understand the self-report assessment forms, or are so severely disabled they cannot comply with the requirements of the study.
6. Individuals with current suicidal risk.
7. Individuals who are legally mandated (e.g., to avoid incarceration, monetary or other penalties, etc.) to participate in substance abuse treatment program.
8. Individuals who are currently receiving any professional treatment (e.g., therapy, medication) for substance abuse problems outside of the current research protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Treatment Engagement | 12 Weeks
  Number of sessions attended
Treatment Completion | 12 Weeks
  Dropout status (completion vs. non-completion)

SECONDARY OUTCOMES:
Cocaine Use | 12 Weeks
  Number of weeks of self-reported abstinence (verified by negative urinary drug screen)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Foltin, Ph.D., Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll, K. M. (1998). A cognitive behavioral approach: treating cocaine addiction. Rockville, MD: National Institute on Drug Abuse.